CLINICAL TRIAL: NCT04791488
Title: Impact of Hyperoxia and Involvement of the Immune System in Diving Accident
Acronym: OXYDIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019PBMD05
Record Dates: First submitted 2020-12-13; First posted 2021-03-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Decompression Sickness
MeSH Terms: conditions — Decompression Sickness | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy individuals (Experimental)
  Interventions: Procedure: Hyperbaric oxygen therapy; Procedure: Diving simulation
- Decompression sickness patients (Experimental)
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy protocol
Procedure: Diving simulation — Hyperbaric chamber diving simulation protocol
  Arms: Healthy individuals

SUMMARY:
The impact of oxygen therapy in many pathologies has been subject of recent work, arguing both favourable and harmful effects. Consequently, one can wonder about the influence of hyperoxic gas mixture during diving on the genesis of decompression sickness, but also about the systematic application of normobaric and hyperbaric oxygen in case of proven decompression sickness.

In mammals, normoxic concentrations have been redefined at 20-100 mbars at the extracellular level and below 10 mbars in the mitochondria.

Under hyperbaric conditions, most of the oxygen being dissolved in blood plasma, a state of hyperoxia is established which escapes the usual delivery and regulation system represented by red blood cells.

The results of our team's previous work suggest a specific effect of diving on the levels of circulating mitochondrial DNA (mtDNA), suggesting cellular destruction linked to hyperoxia/hyperbaria. In fact, our studies, carried out on both animals and human divers, have shown that diving accident leads to an increase in mtDNA levels and an immune reaction through the mobilisation of leukocytes.

The main objective of this study is to compare the influence of oxygen partial pressure levels on the evolution of clinical and biological variables during hyperbaric oxygen therapy sessions in healthy versus injured divers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject with no contraindications to diving OR patient admitted to the hospital for suspicion of a diving accident OR patient admitted to the hospital for hyperbaric oxygen therapy

Exclusion Criteria:

* Contraindication to diving or contraindication to hyperbaric oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of decompression sickness clinical symptoms | Until the end of the oxygen therapy treatment (up to 1 year)
  Decompression sickness clinical symptoms will be assessed through a medical examination after each hyperbaric session.
  Decompression sickness clinical symptoms include: paresthesia, sensory deficit, motor deficit, spinal pain, sphincter disorder and brain injury.
  The evolution of symptoms will be rated as following: total regression, improvement, stabilization, fluctuation or worsening

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Sainte-Anne, Toulon, France

IPD SHARING:
Plan to Share IPD: Undecided